CLINICAL TRIAL: NCT02100332
Title: Prevalence of Comorbidities of COPD in the Exacerbator Phenotype - A Cross Sectional Disease/Condition Focused Observational Study on COPD
Brief Title: A Cross Sectional Disease/Condition Focused Observational Study on Chronic Obstructive Pulmonary Disease (COPD)
Acronym: PREFER
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: RO-2455-402-IT; U1111-1152-9289 (Registry Identifier: WHO (UTN))
Record Dates: First submitted 2014-02-06; First posted 2014-03-31 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic obstructive pulmonary disease: Patients with chronic obstructive pulmonary disease will undergo a single visit with the collection of data from his/her records.

SUMMARY:
The purpose of this study is to establish the prevalence of comorbidities in Italian patients with chronic bronchitis with at least 2 exacerbations per year, and to document the appropriateness of instrumental diagnostic tests, such as spirometry of these patients.

DETAILED DESCRIPTION:
This is an observational study so participants will only take medication that is presently prescribed by their regular healthcare provider. No additional study medication will be administered. This study will enroll patients who have been previously diagnosed with COPD. This study will look at the medical history and other diseases that have been diagnosed in people who also have COPD.

The study will enroll approximately 3000 patients.

This multi-centre trial will be conducted in Italy. The overall time to participate in this study is at a single, regularly scheduled visit at the pulmonologists office. There will not be any follow up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-85, of either gender.
2. Signed informed consent.
3. Known COPD documented by spirometric exams showing fixed non reversible respiratory obstruction.
4. Forced Expired Volume measured after 1 second expiration (FEV-1) < 50% in a previous test (no time limits).
5. Symptoms of chronic bronchitis : chronic productive cough for 3 months at least in each of the 2 years prior to the index visits.
6. On treatment of bronchodilators (no restrictions) for the last 12 months at least.
7. History of at least 2 exacerbations (moderate/severe) in the last 12 months prior to index visit.

Exclusion Criteria:

* None

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD will be enrolled at hospital and pulmonology departments in Italy.
Sampling Method: Probability Sample
Enrollment: 860 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of Comorbidities | Comorbidities captured at the index visit and related to 12 Months Prior to Study Index Visit
  The following comorbidities were accounted for (from the patient records): arterial hypertension, ischemic heart disease, other cardiac disorders, arrhythmia, congestive heart failure, diabetes, metabolic syndrome, known osteoporosis, depression, and chronic renal insufficiency.
Percentage of Participants having Annual Spirometric Tests | 12 months prior and up to the Study Index Visit

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Veruno (Novara), Italy